CLINICAL TRIAL: NCT01029535
Title: Safety and Efficacy of Juvederm® VOLUMA™ for Correction of Mid-face Volume Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VOL-AP01
Record Dates: First submitted 2009-12-08; First posted 2009-12-10 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Mid-face Volume Deficiency

ARMS (1):
- Juvederm® VOLUMA™ (Experimental): Juvederm® VOLUMA™ injected in both sides of face (up to 4 mL per side) at Investigator's discretion to achieve at least a 2-point improvement in the Mid-face Volume Deficit Scale. Participants who completed Week 8 of Phase 1 were eligible to participate in Phase 2 and could receive an additional optional treatment if applicable.
  Interventions: Device: Cross-linked hyaluronic acid gel

INTERVENTIONS:
Device: Cross-linked hyaluronic acid gel — Cross-linked hyaluronic acid gel (Juvederm® VOLUMA™) up to 4 mLs injected in each side of the face.
  Other Names: Juvederm® VOLUMA™

SUMMARY:
This is a prospective, open-label experience study to be conducted at 6 clinical sites in Australia, with the objective to collect efficacy and safety information for Juvederm® VOLUMA™ when used for volumising the mid-face and cheek area.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mild to severe mid-face and cheek volume deficit due to age-related changes, who are likely to improve by at least 2 grades following treatment with the study compound, based on a study-specific scale, as assessed by the study physician

Exclusion Criteria:

* Subjects who have a pre-existing medical condition or who have received any treatments or procedures which may impact on the assessment of the effects of the study compound.
* Subjects with a history of allergies or other side effects to dermal fillers, lidocaine, hyaluronic acid or other component of the study compound.
* Subjects were are pregnant or breast-feeding or who are of child-bearing potential and who are not prepared to practice an adequate form of contraception during the course of the study
* Subjects with a history of alcoholism or drug abuse or dependence

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Sydney, Australia

REFERENCES:
- [Background] Callan P, Goodman GJ, Carlisle I, Liew S, Muzikants P, Scamp T, Halstead MB, Rogers JD. Efficacy and safety of a hyaluronic acid filler in subjects treated for correction of midface volume deficiency: a 24 month study. Clin Cosmet Investig Dermatol. 2013 Mar 20;6:81-9. doi: 10.2147/CCID.S40581. Print 2013. PMID 23687448

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Juvederm® VOLUMA™
Started | 103
Completed | 72
Not Completed | 31
Not completed — Lost to Follow-up | 24
Not completed — Protocol Violation | 2
Not completed — Participant Withdrew Consent | 2
Not completed — Adverse Event | 1
Not completed — Use of Another Treatment | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 103
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 46.7 [29 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥ 1 Point Improvement From Baseline in the Subject's Global Aesthetic Improvement Scale (GAIS) at Week 4
Description: The participant rated their midface appearance compared to Baseline (before treatment) using the 5-point GAIS scale where:-2=much worse to +2=much improved. The percentage of participants +1=improved and +2=much improved is reported.
Time Frame: Baseline, Week 4
Population: Participants from the intent-to-treat (ITT) population, all enrolled participants who received at least one application of VOLUMA™, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 102
percentage of participants | 97.06

2. Primary Outcome: Percentage of Participants With a ≥ 1 Point Improvement From Baseline in the Subject's Global Aesthetic Improvement Scale (GAIS) at Week 8
Description: The participant rated their midface appearance compared to Baseline (before treatment) using the 5-point GAIS scale:-2=much worse to +2=much improved. The percentage of participants +1=improved and +2=much improved is reported.
Time Frame: Baseline, Week 8
Population: Participants from the ITT population, all enrolled participants who received at least one application of VOLUMA™, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 99
percentage of participants | 97.98

3. Primary Outcome: Percentage of Participants With a ≥ 1 Point Improvement From Baseline in the Physician's Global Aesthetic Improvement Scale (GAIS) at Week 4
Description: The physician rated the participant's midface appearance compared to Baseline (before treatment) using the 5-point GAIS scale:-2=much worse to +2=much improved. The percentage of participants +1=improved and +2=much improved is reported.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 102
percentage of participants | 100

4. Primary Outcome: Percentage of Participants With a ≥ 1 Point Improvement From Baseline in the Physician's Global Aesthetic Improvement Scale (GAIS) at Week 8
Description: as for outcome 3
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Number; unit: percentage of particpants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 99
percentage of particpants | 100

5. Primary Outcome: Percentage of Participants a ≥1 Point Improvement From Baseline in the Physician's Mid-face Volume Deficit Scale (MFVDS) at Week 4
Description: The physician determined the degree of midface volume deficiency in each participant, relative to Baseline (before treatment) using the 6-point MFVDS: 0=no facial volume loss to 5=severe volume loss.
Time Frame: Baseline, Week 4
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of particpants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of particpants | 92.23

6. Primary Outcome: Percentage of Participants a ≥ 1 Point Improvement From Baseline in the Physician's Mid-face Volume Deficit Scale (MFVDS) at Week 8
Description: as for outcome 5
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 99
percentage of participants | 95.96

7. Primary Outcome: Percentage of Participants Who Maintained Their Week 8 MFVDS Scores at Week 52
Description: The physician determined the degree of midface volume deficiency in each participant at week 8 and Week 52, relative to before treatment using the 6-point MFVDS: 0-no facial volume loss to 5=severe volume loss. The percentage of participants who are able to maintain their Week 8 score is reported.
Time Frame: Baseline, Week 8, Week 52
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants | 40.8

8. Primary Outcome: Percentage of Participants Who Maintained Their Week 8 MFVDS Scores at Week 78
Description: The physician determined the degree of midface volume deficiency in each participant at week 8 and Week 78, relative to before treatment using the 6-point MFVDS: 0-no facial volume loss to 5=severe volume loss. The percentage of participants who are able to maintain their Week 8 score is reported.
Time Frame: Baseline, Week 8, Week 78
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants | 30.1

9. Primary Outcome: Percentage of Participants Who Maintained Their Week 8 MFVDS Scores at Week 104
Description: The physician determined the degree of midface volume deficiency in each participant at week 8 and Week 104, relative to before treatment using the 6-point MFVDS: 0-no facial volume loss to 5=severe volume loss. The percentage of participants who are able to maintain their Week 8 score is reported.
Time Frame: Baseline, Week 8, Week 104
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants | 38.8

10. Primary Outcome: Percentage of Participants Who Maintained Their Week 8 Subject's GAIS Scores at Week 52
Description: The participant rated their midface appearance compared to before treatment at Week 8 and Week 52 using the 5-point GAIS scale:-2=much worse to +2=much improved. The percentage of participants who are able to maintain their Week 8 score is reported.
Time Frame: Baseline, Week 8, Week 52
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants | 41.7

11. Primary Outcome: Percentage of Participants Who Maintained Their Week 8 Subject's GAIS Scores at Week 78
Description: The participant rated their midface appearance compared to before treatment at Week 8 and Week 78 using the 5-point GAIS scale:-2=much worse to +2=much improved. The percentage of participants who are able to maintain their Week 8 score is reported.
Time Frame: Baseline, Week 8, Week 78
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants | 36.9

12. Primary Outcome: Percentage of Participants Who Maintained Their Week 8 Subject's GAIS Scores at Week 104
Description: The participant rated their midface appearance compared to before treatment at Week 8 and Week 104 using the 5-point GAIS scale:-2=much worse to +2=much improved. The percentage of participants who are able to maintain their Week 8 score is reported.
Time Frame: Baseline, Week 8, Week 104
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants | 36.9

13. Primary Outcome: Percentage of Participants Who Maintained Their Week 8 Physician's GAIS Scores at Week 52
Description: The physician rated the participant's midface appearance compared to before treatment at Week 8 and Week 52 using the 5-point GAIS scale:-2=much worse to +2=much improved. The percentage of participants who are able to maintain their Week 8 score is reported.
Time Frame: Baseline, Week 8, Week 52
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants | 32.0

14. Primary Outcome: Percentage of Participants Who Maintained Their Week 8 Physician's GAIS Scores at Week 78
Description: The physician rated the participant's midface appearance compared to before treatment at Week 8 and Week 78 using the 5-point GAIS scale:-2=much worse to +2=much improved. The percentage of participants who are able to maintain their Week 8 score is reported.
Time Frame: Baseline, Week 8, Week 78
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants | 28.2

15. Primary Outcome: Percentage of Participants Who Maintained Their Week 8 Physician's GAIS Scores at Week 104
Description: The physician rated the participant's midface appearance compared to before treatment at Week 8 and Week 104 using the 5-point GAIS scale:-2=much worse to +2=much improved. The percentage of participants who are able to maintain their Week 8 score is reported.
Time Frame: Baseline, Week 8, Week 104
Population: ITT population included all enrolled participants who received at least one application of VOLUMA™.
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants | 29.1

16. Secondary Outcome: Percentage of Participants With a ≥ 1 Point Improvement From Baseline in the Investigator's Wrinkle Assessment Scale (WAS)
Description: The physician assessed the left side and the right side of the participant's face for severity of nasolabial folds using the 5-point WAS where: 0=no wrinkle to 4=very deep wrinkle.
Time Frame: Baseline, Weeks 4, 8, 52, 78 and 104
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
percentage of participants
  Left Side Week 4 (n=103) | 35.92
  Left Side Week 8 (n=99) | 45.45
  Left Side Week 52 (n=68) | 36.76
  Left Side Week 78 (n=82) | 42.68
  Left Side Week 104 (n=72) | 48.61
  Right Side Week 4 (n=103) | 34.95
  Right Side Week 8 (n=99) | 43.43
  Right Side Week 52 (n=68) | 27.94
  Right Side Week 78 (n=82) | 41.46
  Right Side Week 104 (n=72) | 44.44

17. Secondary Outcome: Change From Baseline in the MFVDS Score
Description: The physician determined the degree of midface volume deficiency in each participant, relative to Baseline (before treatment) using the 6-point MFVDS where: 0=no facial volume loss to 5=severe volume loss. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 52, 78 and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
score on a scale
  Baseline | 3.45 (0.75)
  Change from Baseline at Week 4 | 1.58 (0.83)
  Change from Baseline at Week 8 (n=99) | 2.03 (0.91)
  Change from Baseline at Week 52 (n=68) | 1.68 (0.95)
  Change from Baseline at Week 78 (n=82) | 1.44 (1.04)
  Change from Baseline at Week 104 (n=72) | 1.72 (0.95)

18. Secondary Outcome: Physician Assessment of Global Aesthetic Improvement Score (GAIS)
Description: The physician rated the participant's midface appearance compared to Baseline (before treatment) using the 5-point GAIS scale:-2=much worse to +2=much improved.
Time Frame: Baseline, Weeks 4, 8, 52, 78 and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
score on a scale
  Week 4 (n=102) | 1.35 (0.48)
  Week 8 (n=99) | 1.76 (0.43)
  Week 52 (n=68) | 1.13 (0.81)
  Week 78 (n=82) | 0.85 (0.90)
  Week 104 (n=72) | 1.14 (0.74)

19. Secondary Outcome: Subject's Assessment of Global Aesthetic Improvement Score (GAIS)
Description: The participant rated their midface appearance compared to Baseline (before treatment) using the 5-point GAIS scale:-2=much worse to +2=much improved.
Time Frame: Baseline, Weeks 4, 8, 52, 78 and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
score on a scale
  Week 4 (n=102) | 1.31 (0.52)
  Week 8 (n=99) | 1.55 (0.61)
  Week 52 (n=68) | 1.01 (0.86)
  Week 78 (n=82) | 0.79 (0.94)
  Week 104 (n=72) | 0.97 (0.77)

20. Secondary Outcome: Change From Baseline in the Subject's Self-Perception of Age (SPA)
Description: The participant rated their facial age in years at Baseline and Weeks 4, 8, 52, 78 and 104. A negative change from Baseline indicates an improvement.
Time Frame: Baseline, Weeks 4, 8, 52, 78 and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 103
years
  Change from Baseline at Week 4 (n=101) | -3.03 (3.45)
  Change from Baseline at Week 8 (n=98) | -3.74 (3.99)
  Change from Baseline at Week 52 (n=68) | -3.15 (4.48)
  Change from Baseline at Week 78 (n=82) | -2.88 (4.09)
  Change from Baseline at Week 104 (n=72) | -3.85 (4.01)

21. Secondary Outcome: Percentage of Participants Satisfied or Very Satisfied With the Treatment
Description: Participants rated their satisfaction with treatment using a 5-Point Scale where: 1=very unsatisfied to 5=very satisfied.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Juvederm® VOLUMA™
Number analyzed (Participants) | 99
percentage of participants
  Very Satisfied | 66.7
  Satisfied | 24.2

ADVERSE EVENTS:
Description: 4 Participants did not complete Week 8 of Phase 1 and were not eligible for Phase 2.
Groups:
- Juvederm® VOLUMA™_Phase 1; Juvederm® VOLUMA™_Phase 2: Juvederm® VOLUMA™ injected in both sides of face (up to 4 mL per side) at Investigator's discretion to achieve at least a 2-point improvement in the Mid-face Volume Deficit Scale. Participants who completed Week 8 of Phase 1 were eligible to participate in Phase 2 and could receive an additional optional treatment if applicable.
Arm/Group | Juvederm® VOLUMA™_Phase 1 | Juvederm® VOLUMA™_Phase 2
Serious Adverse Events (participants affected / at risk) | 0/103 | 1/99
Other Adverse Events (participants affected / at risk) | 65/103 | 8/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Juvederm® VOLUMA™_Phase 1 (N=103) | Juvederm® VOLUMA™_Phase 2 (N=99)
Facial swelling (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Juvederm® VOLUMA™_Phase 1 (N=103) | Juvederm® VOLUMA™_Phase 2 (N=99)
Contusion (Skin and subcutaneous tissue disorders) | 49 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 11 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 18 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to release and can embargo communications regarding trial results for a period that is less than or equal to 120 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.